CLINICAL TRIAL: NCT03879148
Title: The Efficacy of Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia Management Following Video Assisted Thoracic Surgery: A Prospective, Randomized Study
Brief Title: Erector Spinae Plane Block for Postoperative Analgesia Management Following Video Assisted Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medipol University Hospital
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer
Keywords: Erector spinae plane block; Video assisted thoracic surgery; Postoperative analgesia
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: randomized prospective study
Who Masked: Outcomes Assessor
Masking Description: Postoperative pain assessment was performed by a anesthetists blinded to the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (Group I) (Active Comparator): The ultrasound (US) guided ESPB was performed under aseptic conditions at the level of T5 vertebrae using the GE Vivid Q® US device. A high frequency 12 MHz linear US probe was covered with a sterile sheath and placed longitudinally 2-3 cm lateral to the T5 transvers process. After visualizing trapezius, rhomboid major, erector spinae muscles superficial to the hyperechoic transverse process shadow respectively, a 22-gauge 50 mm block needle (Braun Stimuplex Ultra 360, Germany) was inserted in a cephalad to caudad direction. Once the needle tip had been placed within the interfacial plane below the erector spinae muscle, 2 mL of saline were injected to confirm the proper injection site, and then a 20 mL dose of 0.25% bupivacaine was injected. Patients received fentanyl via a patient controlled analgesia (PCA) device with a protocol of 2 mL (10 µg/mL) bolus without an infusion dose, 20 min lockout time and 4 hour limit
  Interventions: Other: Erector spinae plane block
- Control group (Group II) (No Intervention): Patients in control group only received fentanyl via a patient controlled analgesia (PCA) device with a protocol of 2 mL (10 µg/mL) bolus without an infusion dose, 20 min lockout time and 4 hour limit.

INTERVENTIONS:
Other: Erector spinae plane block — Erector spinae plane block was performed to the patients under aseptic conditions
  Arms: Erector spinae plane block (Group I)

SUMMARY:
Video assisted thoracic surgery (VATS) has recently been evaluated as the standard surgical procedure for lung surgery. Although VATS is less painful than thoracotomy, patients may feel severe pain during the first hours at postoperative period. Analgesia management is very important for these patients in postoperative period since insufficient analgesia can cause pulmonary complications such as atelectasis, pneumonia and increased oxygen consumption. The ultrasound (US) guided erector spina plane (ESP) block is a novel interfacial plan block defined by Forero et al. at 2016. ESP block provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. In the literature, there is not still any randomized study evaluating ESP block efficiency for postoperative analgesia management after VATS. The aim of this study is to evaluate US-guided ESP block for postoperative analgesia management after VATS.

DETAILED DESCRIPTION:
Postoperative pain after thoracic surgery which is attributed to muscle incision, rib retraction, and intercostal nerve damage may be severe such a degree that it may cause pulmonary complications such as atelectasis, pneumonia and increased oxygen consumption. Because video assisted thoracic surgery (VATS) has some advantages over open thoracotomy such as reduced pain, shoulder dysfunction, early pulmonary impairment, rapid recovery, short hospital stay and low complication risk, it has recently been evaluated as the standard surgical procedure for lung surgery. Although VATS is a less painful procedure than open thoracotomy, patients may still feel severe pain during the first hours at postoperative period. As thoracic epidural analgesia (TEA) is the gold standard analgesic technique after thoracotomy, it is also being used for analgesia management following VATS. Hence TEA has some difficulties in administration and side effects, minimally invasive analgesic techniques are supported for pain management in patients who underwent VATS. The gold standard minimal invasive analgesic technique for VATS is still be questioned. Thoracic paravertebral block (TPVB) has been evaluated as the first step regional analgesia technique after VATS. However, its administration is difficult because of its anatomical proximity to important structures such as the pleura and central neuro-axial system. Therefore it may cause complications such as pneumothorax and neuro-axial injury. The ultrasound (US) guided erector spina plane block (ESPB) - a novel interfacial plan block defined by Forero et al. in 2016 - has the advantage of being away from the pleural and neurological structures, thus the risk of complications is lower. In the literature, case reports about the analgesic effect of ESPB after thoracotomy and VATS has been increasing. However there is no randomized study for VATS yet. In this study, investigators aimed to evaluate the efficacy of US-guided ESPB for postoperative analgesia management following VATS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary lung carcinoma
* Must be undergoing VATS lobectomy under general anesthesia
* Must be in American Society of Anesthesiologists (ASA) classification I-II status

Exclusion Criteria:

* History of bleeding diathesis,
* History of receiving anticoagulant treatment,
* History of local anesthetics or opioid allergy,
* Skin infection at the site of the needle puncture,
* Presence of pregnancy or lactation, and
* Patients who did not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption change is being assessed | Postoperative 1, 2, 4, 8, 16 and 24 hours
  All patients received fentanyl via a patient controlled analgesia (PCA) device.

SECONDARY OUTCOMES:
Postoperative pain scores (Visual analoge score-VAS) is being assessed | Postoperative 1, 2, 4, 8, 16 and 24 hours
  0 = no pain, 10 = the most severe pain felt

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Nagaraja PS, Ragavendran S, Singh NG, Asai O, Bhavya G, Manjunath N, Rajesh K. Comparison of continuous thoracic epidural analgesia with bilateral erector spinae plane block for perioperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):323-327. doi: 10.4103/aca.ACA_16_18. PMID 30052229